CLINICAL TRIAL: NCT05897502
Title: A 34-Week Single-Blind Trial of Explore the Effectors of The Transtheoretical Model on Nutritional Education in Patients on Hemodialysis
Brief Title: Explore the Effectors of The Transtheoretical Model on Nutritional Education in Patients on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liu, Liu-Yin (Other)
Responsible Party: Sponsor-Investigator, Liu, Liu-Yin, Nurse, E-DA Hospital
Organization: E-DA Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: EMRP-112-047
Record Dates: First submitted 2023-05-18; First posted 2023-06-09 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-02

CONDITIONS: End-Stage Kidney Disease; Hyperphosphatemia
Keywords: hemodialysis,nutrition education,The Transtheoretical Model
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The research design explores the evaluation of intervention effectiveness through a parallel group and experimental research design. Intentionally select experimental and control groups. A single blinding design (participants). The experimental group used multi-media education, 20 minutes per session, total 8 courses. The control group received routine education. The Principal investigator explains the research purpose to eligible participant, and signs a consent form. The interviewer conducted data: basic information and nutritional status indicators (mini nutritional assessment scale, dietary knowledge, attitude, behavior scale, simple dietary intake frequency scale) of two groups of hemodialysis patients as the Baseline. After 8-week nutritional education by dialysis nursing staff. Post tests (dietary knowledge, attitude, behavior scale, mini nutritional assessment scale, simple dietary intake frequency scale) were conducted by interviewer at the 3rd, 4th, and 5th months.
Who Masked: Participant
Masking Description: The participant does not know who the intervention group is versus the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the theoretical model nutritional education (Experimental): instruction with multimedia
  Interventions: Behavioral: multimedia education
- control (Placebo Comparator): instruction with traditional paper
  Interventions: Behavioral: multimedia education

INTERVENTIONS:
Behavioral: multimedia education — The experimental group use multimedia education, 20 minute nutrition education courses each time, a total of 8 courses.
  The control group use routine education.
  Other Names: instruction with traditional paper

SUMMARY:
The purpose of this study is to assess the improvement degree of nutritional care program on the nutritional status and eating habits of hemodialysis patients

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written Informed consent will undergo a 1-week screening period to determine eligibility For study entry. At week 0, eligible patients will be assigned to the intervention group and the control group by single-blind manner(participant) with convenience sampling. In the intervention group, the patients were trained in The Transtheoretical Model on nutritional education for 8 weeks. In the control group, the patients were trained in roution nutrition education.

ELIGIBILITY:
Inclusion Criteria:

1. the biochemical value ≥ 5.5 mg/dl or albumin value<3.8g/dL
2. BMI<23kg/m2
3. Unexpected weight loss.
4. Must be able to swallow tablets

Exclusion Criteria:

1. Clinical diagnosis of Alzheimer's Disease
2. Malignant tumors, gastrointestinal cachexia, and catheterization

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Biochemical value (Albumine) at the third month | Baseline and the third month
  Biochemical value (Albumine) is a validated to assess the nutritional status of hemodialysis, less than 3.8gm/dl is considered malnutrition
Change from Baseline in Biochemical value (Albumine) at the fourth month | Baseline and the fourth month
  Biochemical value (Albumine) is a validated to assess the nutritional status of hemodialysis, less than 3.8gm/dl is considered malnutrition
Change from Baseline in Biochemical value (Albumine) at the sixth month | Baseline and the sixth month
  Biochemical value (Albumine) is a validated to assess the nutritional status of hemodialysis, less than 3.8gm/dl is considered malnutrition
Change from Baseline in Biochemical value( normalized protein catabolic rate) at the third month | Baseline and the third month
  Biochemical value( normalized protein catabolic rate) is a validated to assess the nutritional status of hemodialysis, normal value greater than 1.2gm/day/k
Change from Baseline in Biochemical value( normalized protein catabolic rate) at the fourth month | Baseline and the fourth month
  Biochemical value( normalized protein catabolic rate) is a validated to assess the nutritional status of hemodialysis, normal value greater than 1.2gm/day/k
Change from Baseline in Biochemical value( normalized protein catabolic rate) at the sixth month | Baseline and the sitxth month
  Biochemical value( normalized protein catabolic rate) is a validated to assess the nutritional status of hemodialysis, normal value greater than 1.2gm/day/k
Change from Baseline in Biochemical value(cholesterol )at the third month | Baseline and the third month
  Biochemical value( cholesterol) is a validated to assess the nutritional status of hemodialysis, less than 100mg/dl is considered malnutrition
Change from Baseline in Biochemical value(cholesterol )at the fourth month | Baseline and the fourth month
  Biochemical value( cholesterol) is a validated to assess the nutritional status of hemodialysis, less than 100mg/dl is considered malnutrition
Change from Baseline in Biochemical value(cholesterol )at the sixth month | Baseline and and the sixth month
  Biochemical value( cholesterol) is a validated to assess the nutritional status of hemodialysis, less than 100mg/dl is considered malnutrition
Change from Baseline in Biochemical value(creatine)at the third month | Baseline and the third month
  Biochemical value(creatine) is a validated to assess the nutritional status of hemodialysis, less than 8-10 mg/dl before hemodialysis indicates malnutrition
Change from Baseline in Biochemical value(creatine) at the fourth month | Baseline and the fourth month
  Biochemical value(creatine) is a validated to assess the nutritional status of hemodialysis, less than 8-10 mg/dl before hemodialysis indicates malnutrition
Change from Baseline in Biochemical value(creatine) at the sixth month | Baseline and the sixth month
  Biochemical value(creatine) is a validated to assess the nutritional status of hemodialysis, less than 8-10 mg/dl before hemodialysis indicates malnutrition
Change from Baseline in Biochemical value( Phosphate) at the third month | Baseline and the third month
  Biochemical value(Phosphate) is a validated to assess the nutritional status of hemodialysis, normal value is 2.7-4.5 mg/dL
Change from Baseline in Biochemical value( Phosphate) at the fourth month | Baseline and the fourth month
  Biochemical value(Phosphate) is a validated to assess the nutritional status of hemodialysis, normal value is 2.7-4.5 mg/dL
Change from Baseline in Biochemical value( Phosphate) at the sixth month | Baseline and the sixth month
  Biochemical value(Phosphate) is a validated to assess the nutritional status of hemodialysis, normal value is 2.7-4.5 mg/dL
Change from Baseline in body measurement ( Hand grip strength ) at the third month | Baseline and the third month
  Hand grip strength is a validated to assess the nutritional status of hemodialysis, male ≤ 30 kilograms, female ≤ 20 kilograms, indicating a risk of frailty
Change from Baseline in body measurement ( Hand grip strength ) at the fourth month | Baseline and the fourth month
  Hand grip strength is a validated to assess the nutritional status of hemodialysis, male ≤ 30 kilograms, female ≤ 20 kilograms, indicating a risk of frailty
Change from Baseline in body measurement ( Hand grip strength ) at the sixth month | Baseline and the sixth month
  Hand grip strength is a validated to assess the nutritional status of hemodialysis, male ≤ 30 kilograms, female ≤ 20 kilograms, indicating a risk of frailty
Change from Baseline in (Mini Nutritional Assessment-Short Form, MNA-SF) at the third month | Baseline and the third month
  (Mini Nutritional Assessment-Short Form, MNA-SF) is a validated self-reported instrument to assess the nutritional status of hemodialysis,Out of 14 points. ≤11 points malnutrition risk. ≤7 points malnutrition.
Change from Baseline in (Mini Nutritional Assessment-Short Form, MNA-SF) at the fourth month | Baseline and the fourth month
  (Mini Nutritional Assessment-Short Form, MNA-SF) is a validated self-reported instrument to assess the nutritional status of hemodialysis,Out of 14 points. ≤11 points malnutrition risk. ≤7 points malnutrition.
Change from Baseline in (Mini Nutritional Assessment-Short Form, MNA-SF) at the sixth month | Baseline and the six month
  (Mini Nutritional Assessment-Short Form, MNA-SF) is a validated self-reported instrument to assess the nutritional status of hemodialysis,Out of 14 points. ≤11 points malnutrition risk. ≤7 points malnutrition.

SECONDARY OUTCOMES:
Change from Baseline in the diet of knowledge form at the third month | Baseline and the third month
  The diet of knowledge form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 10 points. The higher the score, the positive performance on healthy diet knowledge
Change from Baseline in the diet of knowledge form at the fourth month | Baseline and the fourth month
  The diet of knowledge form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 10 points. The higher the score, the positive performance on healthy diet knowledge
Change from Baseline in the diet of knowledge form at the sixth month | Baseline and the sixth month
  The diet of knowledge form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 10 points. The higher the score, the positive performance on healthy diet knowledge
Change from Baseline in the diet of attitude form at the third month | Baseline and the third month
  The diet of attitude form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 20 points. A higher score indicates a positive attitude towards healthy eating
Change from Baseline in the diet of attitude form at the fourth month | Baseline and the fourth month
  The diet of attitude form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 20 points. A higher score indicates a positive attitude towards healthy eating
Change from Baseline in the diet of attitude form at the sixth month | Baseline and the sixth month
  The diet of attitude form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 20 points. A higher score indicates a positive attitude towards healthy eating
Change from Baseline in the diet of behavior form at the third month | Baseline and the third month
  The diet of behavior form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 20 points. A higher score indicates a positive performance on healthy eating behavior
Change from Baseline in the diet of behavior form at the fourth month | Baseline and the fourth month
  The diet of behavior form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 20 points. A higher score indicates a positive performance on healthy eating behavior
Change from Baseline in the diet of behavior form at the sixth month | Baseline and the sixth month
  The diet of behavior form is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 20 points. A higher score indicates a positive performance on healthy eating behavior
Change from Baseline in the high phosphorus food frequency questionnaire at the third month | Baseline and the third month
  The high phosphorus food frequency questionnaire is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 42. The higher the score, the negative the frequency of food intake with high phosphorus.
Change from Baseline in the high phosphorus food frequency questionnaire at the fourth month | Baseline and the fourth month
  The high phosphorus food frequency questionnaire is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 42. The higher the score, the negative the frequency of food intake with high phosphorus.
Change from Baseline in the high phosphorus food frequency questionnaire at the sixth month | Baseline and the sixth month
  The high phosphorus food frequency questionnaire is a validated self-reported instrument to assess the eating habits of hemodialysis patients,The full score is 42. The higher the score, the negative the frequency of food intake with high phosphorus.
Change from Baseline in the six major food frequency questionnaire at the third month | Baseline and the third month
  The six major food frequency questionnaire is a validated self-reported instrument to assess the eating habits of hemodialysis patients,Full score is 12 points. A higher score indicates a balanced performance on the six major food intake frequencies
Change from Baseline in the six major food frequency questionnaire at the fourth month | Baseline and the fourth month
  The six major food frequency questionnaire is a validated self-reported instrument to assess the eating habits of hemodialysis patients,Full score is 12 points. A higher score indicates a balanced performance on the six major food intake frequencies
Change from Baseline in the six major food frequency questionnaire at the sixth month | Baseline and the sixth month
  The six major food frequency questionnaire is a validated self-reported instrument to assess the eating habits of hemodialysis patients,Full score is 12 points. A higher score indicates a balanced performance on the six major food intake frequencies

CONTACTS AND LOCATIONS:
Overall Officials: liu-yin Liu, Principal Investigator — The Nursing department of EDAHospital
Locations (1):
- Liu liu.yin, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Based on the privacy and confidentiality factors of the subjects' personal data

REFERENCES:
- [Result] Karavetian M, Elzein H, Rizk R, Jibai R, de Vries N. Nutritional education for management of osteodystrophy: Impact on serum phosphorus, quality of life, and malnutrition. Hemodial Int. 2016 Jul;20(3):432-40. doi: 10.1111/hdi.12405. Epub 2016 Feb 3. PMID 26843138
- See also: I will refer to the food composition analysis in the materials, and the part about phosphorus and protein will be the basis of the research. — https://consumer.fda.gov.tw